CLINICAL TRIAL: NCT05182996
Title: Perceptions and Barriers About Cessation of Smoking Among IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, YooJin Lee, Assistant Professor, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-07-037
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Smoking; Inflammatory Bowel Diseases
MeSH Terms: conditions — Smoking; Inflammatory Bowel Diseases | interventions — Smoking Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- smoking education (Other): smoking education
  Interventions: Behavioral: smoking education

INTERVENTIONS:
Behavioral: smoking education — Educate on the relationship between inflammatory bowel disease and smoking and the necessity and importance of quitting smoking.

SUMMARY:
This study will investigate the perception of the relationship between smoking and inflammatory bowel disease by surveying inflammatory bowel disease patients. Afterward, the relationship between smoking and inflammatory bowel disease will be explained, and the smoking cessation rate will be investigated three months later.

DETAILED DESCRIPTION:
A survey is conducted on patients with inflammatory bowel disease (IBD). Current smoking status, daily smoking amount, smoking period, perception of smoking effect on the induction of Crohn's disease (CD) or ulcerative colitis (UC), and perception of the effect of smoking on the course of CD or UC were investigated. Moreover, the intention to quit smoking is investigated. After the survey, information on the effects of smoking on CD or IBD is provided, and smoking cessation education is provided. After three months, the patients' smoking behavior was investigated, and the smoking cessation rate was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with inflammatory bowel disease or newly diagnosed with inflammatory bowel disease

Exclusion Criteria:

* Those who do not agree to the survey or smoking cessation education

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
smoking cessation rate | 3 month later
  Percentage of smokers who succeeded in quitting smoking

CONTACTS AND LOCATIONS:
Locations (1):
- KeimyungUniversity, Daegu, Jung-gu, South Korea